CLINICAL TRIAL: NCT07268729
Title: Investigation of Pathogenic Gut Microbiota Patterns in Anxiety, Depression and Panic Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: University of Toronto (Other)
Collaborators: MedBliss Research Network (Unknown)
Responsible Party: Principal Investigator, Hassan Kattan, Principal Investigator, University of Toronto
Other Study IDs: Pro00084759
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Panic Disorder; Mood Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Mood Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients under ongoing treatment: Participants in this group are adults currently receiving ongoing treatment for anxiety, depression, or panic disorder. Treatment may include prescribed medication, psychotherapy, or other clinician-supervised care. These participants will complete the same baseline psychological assessments and stool microbiome testing as the other cohorts. Their data will help evaluate how existing treatments may influence gut microbiome composition and mental-health outcomes over time.
  Interventions: Diagnostic Test: H pylori stool test; Diagnostic Test: Bacterial stool analysis
- Healthy controls with no psychiatric history: Participants in this group are healthy adults with no self-reported or clinically diagnosed history of psychiatric or neurological disorders. They will complete the same baseline assessments and biological sample collection (including stool microbiome testing) as the clinical cohort, but will not receive any treatment or individualized intervention. Their data will serve as a comparison reference to help identify microbiome and biomarker patterns associated with anxiety and depression.
  Interventions: Diagnostic Test: H pylori stool test; Diagnostic Test: Bacterial stool analysis
- Patients with clinically confirmed anxiety, depression, and panic disorder.: Participants in this cohort are adults with a current, clinically confirmed diagnosis of anxiety disorder, depressive disorder, or panic disorder. Each participant will provide baseline psychological assessments and biological samples, including stool microbiome testing. Based on their results, they may receive individualized lifestyle or dietary recommendations under physician supervision. Participants will be followed over time to evaluate changes in mood, stress, and biological markers related to mental-health outcomes.
  Interventions: Diagnostic Test: H pylori stool test; Diagnostic Test: Bacterial stool analysis

INTERVENTIONS:
Diagnostic Test: H pylori stool test — Participants will provide a stool sample for noninvasive testing to detect the presence of Helicobacter pylori bacteria. The test will be performed using a validated laboratory assay that identifies H. pylori antigens in stool. Results will be used to assess potential associations between H. pylori infection, gut microbiome composition, and symptoms of anxiety or depression. The test is diagnostic only and does not involve administration of any drug or treatment.
Diagnostic Test: Bacterial stool analysis — Participants will provide stool samples for microbiome sequencing using a validated laboratory assay. The analysis will characterize bacterial taxa within the gut microbiome and identify potential pathogenic species. Sequencing results will be correlated with psychological assessments and clinical measures to investigate relationships between gut microbial composition and symptoms of anxiety, depression, and panic disorder.

SUMMARY:
This study aims to investigate the etiology of anxiety, depression, and panic disorders, providing new evidence and insights into the root causes and effective treatments, potentially offering a novel approach to achieving complete recovery.

DETAILED DESCRIPTION:
Background: Anxiety, depression and panic disorders are among the most prevalent mental health conditions globally, affecting millions and imposing a substantial burden on individuals, families, and healthcare systems. These disorders often manifest through recurrent, severe episodes of anxiety and fear, frequently accompanied by physical symptoms such as palpitations, chest pain, and dizziness, which can lead to significant functional impairment and diminished quality of life. While current treatment options include pharmacotherapy and cognitive-behavioral therapy, response rates vary, and many patients experience residual symptoms or adverse effects, leading to high rates of treatment discontinuation. Furthermore, the growing recognition of treatment-resistant anxiety, depression and panic disorders highlights an urgent need for innovative, evidence-based therapies that provide sustained relief without compromising safety.

Introduction Anxiety, depression and panic disorders are pervasive and debilitating chronic mental health conditions, affecting approximately 20% of the global population over a lifetime. Characterized by episodes of intense fear and physical symptoms such as heart palpitations, shortness of breath, and dizziness, these disorders can severely impact daily functioning, interpersonal relationships, and overall quality of life. Individuals with these conditions are also at increased risk for comorbidities including depression, substance use disorders, and cardiovascular disease, further complicating their clinical profile and necessitating more comprehensive treatment strategies.

Despite the availability of pharmacotherapy, such as selective serotonin reuptake inhibitors (SSRIs) and benzodiazepines, alongside cognitive-behavioral therapy (CBT), there remain substantial challenges in achieving and maintaining symptom relief. Response rates vary widely, and a significant proportion of patients experience partial or inadequate relief, with some exhibiting treatment-resistant symptoms. Moreover, pharmacological treatments can be associated with side effects like weight gain, fatigue, and cognitive impairment, which may lead to discontinuation or non-adherence. These limitations highlight a critical need for alternative or adjunctive interventions that can provide more effective, sustainable, and safer outcomes.

This trial was therefore designed to assess the prevalence of pathogenic gut bacteria among patients with anxiety, depression, and panic disorder compared to healthy controls.

Objective: This study aims to investigate the etiology of anxiety, depression, and panic disorders, providing new evidence and insights into the root causes, potentially offering a novel approach to these conditions..

Findings from this study are anticipated to advance clinical understanding and treatment options for anxiety, depression and panic disorders, providing a potentially more effective approach and that provide lasting relief for patients struggling with these conditions.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 18-65 years.

  * Either of the following:

    1. Diagnosed with anxiety, depression, or panic disorder according to DSM-5 criteria, regardless of current treatment status.
    2. Healthy individuals with no history of psychiatric disorders (control group).
  * Able to provide informed consent and stool sample.

Exclusion Criteria:

* • Diagnosis of psychotic disorders or neurocognitive conditions.

  * Use of systemic antibiotics or antifungals within the past 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult males and females aged 18 to 65 recruited from the general population and outpatient mental health clinics. Participants will include individuals with clinically confirmed anxiety, depression, or panic disorder, as well as healthy control subjects with no psychiatric history. The study will aim to include participants from diverse ethnic and cultural backgrounds to ensure broad representation of the population.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Presence of pathogenic gut bacteria | Day 10 Upon receipt of stool analysis results
  The presence of pathogenic bacterial species will be identified through microbiome sequencing of stool samples using a validated laboratory assay. Sequencing data will be analyzed to detect and quantify bacterial taxa associated with dysbiosis and pathogenicity within the gut microbiome. The primary outcome will be defined as the detection of one or more bacterial pathogens meeting pre-specified taxonomic or functional criteria.

SECONDARY OUTCOMES:
Symptom reduction, and eradication. | Day 0 (baseline), Day 24 (post-eradication reassessment), and Day 30 (post-eradication reassessment)
  Changes in psychological symptom severity will be assessed using validated clinical instruments for anxiety, depression, and panic disorder. Composite symptom scores will be calculated and compared with baseline values to evaluate reductions in symptom severity over time. Correlations between the eradication of pathogenic gut bacteria and improvements in psychological symptoms will also be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- MedBliss Research Network, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy considerations and data governance restrictions related to identifiable microbiome and psychological data. Summary results and aggregated findings will be made publicly available through publication and ClinicalTrials.gov reporting.